CLINICAL TRIAL: NCT04327557
Title: Pilot Study on Effectiveness of Childbirth Education
Brief Title: Childbirth Education Pilot Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-1575; A271000 (Other: UW Madison); SOHE/GENERAL ADMINISTRATION (Other: UW Madison); Protocol Version 2/3/2020 (Other: UW Madison)
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either MBCP childbirth education course or a non-MBCP childbirth course to look at effects of different types of childbirth education.
Who Masked: Participant
Masking Description: There is no mention of MBCP as an option for childbirth education classes in the consent form or recruitment materials, but participants who are randomized to the MBCP group do find out that they are in the MBCP group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCP Childbirth Education Course (Experimental): This arm will undergo the 9-week MBCP course.
  Interventions: Behavioral: MBCP Childbirth Education Course
- Non-MBCP Childbirth Education Course (Active Comparator): This arm will undergo the TAU (treatment as usual) childbirth education course (one that does not have a huge mindfulness component).
  Interventions: Behavioral: Non-MBCP Childbirth Education Course

INTERVENTIONS:
Behavioral: MBCP Childbirth Education Course — The MBCP program is a fully manualized childbirth and parenting preparation course. Developed in 1998 in a clinical context, MBCP is an enhanced version of the Mindfulness Based Stress Reduction (MBSR) program tailored for addressing the concerns of pregnancy and early parenting. Through MBCP, pregnant women and their partners learn mindfulness skills for coping with the anxiety and stress of pregnancy and parenting, and the pain and fear of childbirth. They are given explicit instruction in skills for cultivating positive emotion and developing mindful, sensitive parenting. MBCP groups meet weekly for 9 weeks, with a retreat day between weeks 6 and 7.
  Arms: MBCP Childbirth Education Course
Behavioral: Non-MBCP Childbirth Education Course — TAU control participants will undergo standard (real-world) hospital- or community-based childbirth education that does not have a mindfulness focus. They will be able to choose whichever class they want from the list. If they prefer a class that is not on the list, then study staff will obtain the syllabus for that class to check whether there is a mindfulness component.
  Arms: Non-MBCP Childbirth Education Course

SUMMARY:
This study aims to investigate the effects of mindfulness training on prenatal maternal anxiety using a randomized controlled trial (RCT). An RCT of mindfulness training for prenatal anxiety has distinct clinical and scientific advantages.

The investigators will use the Mindfulness-Based Childbirth and Parenting (MBCP) intervention in this study to build on previous findings by focusing on anxiety in pregnancy while also teaching mindfulness skills shown to promote positive childbirth appraisals and sensitive parenting through mindful parenting skills that have been shown to be linked to maternal-infant stress physiology in other work.

This study will enroll pregnant women with elevated anxiety (N = 60) who will be randomly assigned to the MBCP condition (n = 30) or an active control condition (a treatment as usual (TAU) condition; n = 30) which is a standard childbirth education class. Mothers will be assessed pre- and post-intervention and postpartum. Infant multi-modal neuroimaging will occur at age 1 month, at home questionnaire follow-up will occur at age 3 months, and a behavioral observation of parenting and child social-emotional functioning will occur at age 12 months. The hypothesis is that there will be greater benefits from MBCP relative to TAU controls, and enhanced connectivity between the amygdala and relevant cortico-limbic areas in from MBCP relative to TAU controls.

DETAILED DESCRIPTION:
Baseline (Pre-Class) Visit : Once study eligibility has been confirmed, the participant will come to the lab for an in-person visit. If they choose to continue in the study after reading and signing the consent form, they will complete a series of questionnaires and collect saliva samples at home.

Childbirth Education Intervention: The participant will be randomly assigned to one of two childbirth and parenting education groups (either the MBCP course offered at UW Health or a TAU course). Participants in the TAU group will be provided options of courses to select. Courses may last up to 9 weeks long. The course is provided as part of the study. Participants are asked to complete the course before the 37th week of pregnancy.

Post-Intervention (Post-Class) Visit: After completing the childbirth and parenting education course, the participant will complete a series of questionnaires and collect another set of saliva samples. This can happen in person or remotely.

1-Month Follow-Up Visit: One month after birth, the participant and their child will come to the lab for an MRI scan of the child's brain while he or she sleeps as well as complete another series of questionnaires.

3-Month Follow-Up Visit: Three months after birth, the participant will complete a series of questionnaires.

12-Month Follow-Up Visit: Twelve months after birth, the participant and their child will come to the lab for one final visit to do a behavioral assessment as well as complete a final series of questionnaires.

ELIGIBILITY:
Maternal Inclusion Criteria:

* A score on the Penn State Worry Questionnaire (PSWQ) of 50 or greater
* Nulliparous and expecting a healthy (i.e., normal/low medical risk), singleton pregnancy
* No more than 28 weeks gestation at time of enrollment (to allow time to complete the intervention before 37 weeks)
* Comfortable reading, writing, and conversing in English.
* Available and able to enroll in the MBCP class

Infant Inclusion Criteria:

* Born to a mother participating in the study

Maternal Exclusion Criteria:

* Severe medical conditions that would compromise the pregnancy (e.g., pre-eclampsia, severe hyperthyroidism);
* Current or past bipolar disorder, schizophrenia, or post-traumatic stress disorder (PTSD);
* Active psychopharmacological treatment (current or in the past 6 months).
* Formal mindfulness meditation practice or long-term yoga practice
* Significant injuries, illness or surgery that may impair parent-child interaction (e.g., traumatic brain injury) or that is unstably treated.
* HIV or AIDS
* Cancer in the past year
* Major Autoimmune Disease
* Infection while pregnant such as Toxoplasmosis, Rubella, Cytomegalovirus (CMV) infection, Herpes Simplex Virus (HSV), Syphilis
* Prior childbirth

Infant Exclusion Criteria:

* Major neurosensory impairment: legally blind or coloboma
* Isoimmunization
* Severe jaundice
* Facial cleft
* Abnormal heart rate: ECG >180 or <80

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Maternal Stress Physiology as Measured by Change in Slope for Salivary Cortisol from Pre-Class to Post-Class Phase | At pre-class and post-class phases approximately within a 12 week window
  Salivary cortisol will be collected at home 3 times per day (upon waking, 40 minutes post waking, and before bed) for 3 days to provide measures of cortisol diurnal rhythm. Kits will be sent home for participants to use. Mean diurnal cortisol will be reported for each time point (waking, 40 minutes post waking, and before bed). Then the change in slope from the pre-class samples to the post-class samples will be investigated. Collection will occur within 1 week of completion of pre-class questionnaires and within 1 week after completion of the childbirth education course and post-class questionnaires.
Change in Anxiety Levels as Measured by the State Trait Anxiety Inventory-X2 (STAI-X2) | Up to 12 months post birth
  Change in anxiety level will be explored using the STAI-X2 scale which will also be used to compare the Mindfulness-Based Childbirth and Parenting (MBCP) group to the Treatment as usual (TAU) group.
  The STAI-X2 is a 20-item self-report questionnaire designed to evaluate anxiety in adults. Ratings are on a 4-point scale: 0-Not at all, 1-Somewhat, 2-Moderately so, 3-Very much so. Total possible range of scores is 0-60, higher scores reflect greater symptomatology of anxiety. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Depression Levels as Measured by the Edinburgh Postnatal Depression Scale (EPDS) | Up to 12 months post birth
  Change in depression level will be explored using the EPDS which will also be used to compare the MBCP group to the TAU group.
  The EPDS is a 10-item self-report questionnaire that can indicate symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child. Ratings are on a 4-point scale. Total possible range of scores is 0-30, higher scores reflect greater symptomatology of depression. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Depression Levels as Measured by the Center for Epidemiologic Studies Depression (CESD) Scale | Up to 12 months post birth
  Change in depression level will be explored by using the CESD scale which will also be used to compare the MBCP group to the TAU group.
  The CESD scale is a 20-item self-report questionnaire comprising six scales reflecting major facets of depression: depressed mood, feelings of guilt and worthlessness, feelings of helplessness and hopelessness, psychomotor retardation, loss of appetite, and sleep disturbance. Ratings are on a 4-point scale. Total possible range of scores is 0-60, higher scores reflect greater symptomatology of depression. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Positive and Negative Emotions as Measured by the Positive And Negative Affect Scale (PANAS) | Up to 12 months post birth
  Change in positive and negative emotions will be explored using the PANAS which will also be used to compare the MBCP group to the TAU group.
  The PANAS is a self-report questionnaire that is split into two segments, or mood scales, of 10-items each. One scale measures a person's positive emotion and the other measures negative emotion. Ratings are on a 5-point scale. Total possible range of scores in the positive segment is 10-50 with higher scores indicating higher positive mood. Total possible range of scores in the negative segment is 10-50 with higher scores indicating higher negative mood. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Emotional State as Measured by the Differential Emotions Scale (DES) | Up to 12 months post birth
  Emotional state will be explored using the DES which will also be used to compare the MCBP group to the TAU group.
  The DES is a 19-item self-report questionnaire that divides the individual's description of emotion experience into validated, discrete categories of emotion. The DES was formulated to gauge the emotional state of individuals at that specific point in time when they are responding to the instrument. Ratings are on a 5-point scale. Total possible range of scores in the positive segment is 0-40 with higher scores indicating higher positive mood. Total possible range of scores in the negative segment is 0-36 with higher scores indicating higher negative mood. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Mindfulness Levels as Measured by the Five Facet Mindfulness Questionnaire (FFMQ) | Up to 12 months post birth
  Elements of mindfulness will be explored using the FFMQ which will also be used to compare the MBCP group to the TAU group.
  The FFMQ is a 39-item self-report questionnaire consisting of five subscales (observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience). Ratings are on a 5-point scale. Total possible range of scores is 8-40 for each of the subscales except non-reactivity to inner experience which has a total possible range of 7-35 with higher scores indicating higher elements of mindfulness. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Worry Levels as Measured by the Penn State Worry Questionnaire (PSWQ) | Up to 12 months post birth
  Change in worry level will be explored using the PSWQ which will also be used to compare the MBCP group to the TAU group.
  The PSWQ is a 16-item self-report questionnaire that is designed to measure worry. The items on the scale assess the occurrence, intrusiveness, pervasiveness, and other characterizing features of an individual's experience with worry. The scale has been shown to identify worry, over and above anxiety and depression. Ratings are on a 5-point scale: 1-Not at all typical of me to 5-Very typical of me. Total possible range of scores is 16-80 with 16-39 indicating low worry, 40-59 moderate worry, and 60-80 high worry. This outcome is assessed at all phases except pre-class (screening, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Infant Emotion Regulation as Measured by the Infant Behavior Questionnaire-Revised (IBQ-R) | At 3 month and 12 month post birth
  Infant emotion regulation will be explored using the IBQ-R which will also be used to compare the MBCP group to the TAU group.
  The IBQ-R is a 191-item self-report questionnaire which assesses 14 domains of infant temperament (activity level, distress to limitations, approach, fear, duration of orienting, smiling and laughter, vocal reactivity, sadness, perceptual sensitivity, high-intensity pleasure, low-intensity pleasure, cuddliness, soothability, and falling reactivity/rate of recovery from distress). The items on the IBQ-R ask parents to rate the frequency of specific temperament-related behaviors observed over the past week (or 2 weeks for some items). Ratings are on a 7-point scale: 1-Never to 7-Always. This outcome is assessed at the 3 month and 12 month follow-up phases.
Change in Parenting Stress Levels as Measured by the Parenting Stress Index-Short Form (PSI-SF) | At 1 month, 3 month and 12 month post birth
  Change in parenting stress level will be explored using the PSI-SF which will also be used to compare the MBCP group to the TAU group.
  The PSI-SF is a 31-item self-report questionnaire that is a direct derivative of the PSI full-length test for parents of children 12 years and younger. The PSI-SF yields a total stress score from three scales: parental distress, parent-child dysfunctional interaction, and difficult child. Ratings are on a 5-point scale: 1-strongly disagree to 5-strongly agree. Total possible range of scores is 31-155 with higher scores indicating higher stress. This outcome is assessed at the 1 month, 3 month, and 12 month follow-up phases.
Change in Parenting Competence Levels as Measured by the Parenting Sense of Competence Scale (PSC) | At 1 month, 3 month and 12 month post birth
  Change in parenting competence level will be explored using the PSC which will also be used to compare the MBCP group to the TAU group.
  The PSC scale is a 17-item self-report questionnaire that measures parental competence on two dimensions: satisfaction and efficacy. The 9-item satisfaction dimension examines the parents' anxiety, motivation and frustration, while the 8-item efficacy dimension looks at the parents' competence, capability levels, and problem-solving abilities in their parental role. Ratings are on a 6-point scale: 1-strongly agree to 6-strongly disagree. Items 2, 3, 4, 5, 8, 9, 12, 14, and 16 are reverse scored. Higher scores indicate higher parenting sense of competency. This outcome is assessed at the 1 month, 3 month, and 12 month follow-up phases.
Change in Compassion Levels as Measured by the Compassion Scale (CS) | Up to 12 months post birth
  Change in compassion level will be explored using the CS which will also be used to compare the MBCP group to the TAU group.
  The CS is a 16-item self-report questionnaire comprised of 4 subscales: kindness, common humanity, mindfulness, and indifference. Ratings are on a 5-point scale: 1-almost never to 5-almost always. Total possible range of scores is 16-80 with higher scores indicating higher compassion. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Self-Compassion Levels as Measured by the Self-Compassion Scale-Short Form (SCS-SF) | Up to 12 months post birth
  Change in self-compassion level will be explored using the SCS-SF which will also be used to compare the MBCP group to the TAU group.
  The SCS-SF is a 12-item self-report questionnaire that is a direct derivative of the full-length SCS. It is comprised of 6 subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identified. Participants rate how they typically act towards themselves in difficult times. Ratings are on a 5-point scale: 1-almost never to 5-almost always. To compute a total self-compassion score, reverse score the negative subscale items - self-judgment, isolation, and over-identification and then compute a total mean. Higher scores indicate higher self-compassion. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Antenatal Attachment Levels as Measured by the Maternal Antenatal Attachment Scale (MAAS) | At pre-class and post-class phases approximately within a 12 week window
  Change in antenatal attachment level will be explored using the MAAS which will also be used to compare the MBCP group to the TAU group.
  The MAAS is a 19-item self-report questionnaire comprised of 3 subscales: quality of attachment, absence of hostility, and pleasure in interaction. Ratings are on a 5-point scale. Total possible range of scores is 19-95. Items 1, 3, 5, 6, 7, 9, 10, 12, 15, 16, and 18 are reverse scored. This outcome is assessed at pre-class and post-class phases.
Change in Postnatal Attachment Levels as Measured by the Maternal Postnatal Attachment Scale (MPAS) | At 1 month, 3 month and 12 month post birth
  Change in postnatal attachment level will be explored using the MPAS which will also be used to compare the MBCP group to the TAU group.
  The MPAS is a 19-item self-report questionnaire comprised of 2 subscales: quality of attachment and time spent in attachment (or intensity of preoccupation). Ratings are on a 5-point scale. Total possible range of scores is 19-95. Items 7, 8, 9, 10, 11, 12, 13, and 14 are reverse scored. This outcome is assessed at the 1 month, 3 month, and 12 month follow-up phases.
Change in Parental Mindfulness Levels as Measured by the Interpersonal Mindfulness in Parenting (IM-P) Questionnaire | At 1 month, 3 month and 12 month post birth
  Change in parental mindfulness level will be explored using the IM-P which will also be used to compare the MBCP group to the TAU group.
  The IM-P is a 10-item self-report questionnaire that measures mindful parenting. Ratings are on a 5-point scale: 1-Never true to 5-Always true. Total possible range of scores is 10-50. Items 1, 5, 9, and 10 are reverse scored. Higher scores indicate higher parental mindfulness. This outcome is assessed at the 1 month, 3 month, and 12 month follow-up phases.
Physical Activity Levels as Measured by the International Physical Activity Questionnaire-Long (IPAQ-Long) | At 1 month, 3 month and 12 month post birth
  Physical activity level will be explored using the IPAQ-Long which will also be used to compare the MBCP group to the TAU group.
  The IPAQ-Long is a 27-item self-report questionnaire comprised of 5 activity domains. A continuous score is expressed as Metabolic Equivalent (MET)-min per week: MET level x minutes of activity x events per week. This outcome is assessed at the 1 month, 3 month, and 12 month follow-up phases.
Change in Sleep Quality Levels as Measured by the General Sleep Disturbance Scale (GSDS) | Up to 12 months post birth
  Change in sleep quality level will be explored using the GSDS which will also be used to compare the MBCP group to the TAU group.
  The GSDS is a 21-item self-report questionnaire initially designed to evaluate the incidence and nature of sleep disturbances in employed women. Questions pertain to a variety of general sleep issues: problems initiating sleep, waking up during sleep, waking too early from sleep, quality of sleep, quantity of sleep, fatigue and alertness at work, and the use of substances to induce sleep. Ratings are on a 6-point scale. Total possible range of scores is 0-147. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Pregnancy Substance Use as Measured by Retrospective Substance Use (RSU) | At post-class phase within a 1 week window
  Pregnancy substance will be explored using the RSU which will also be used to compare the MBCP group to the TAU group.
  The RSU is an 8-item self-report questionnaire asking participant to retrospectively answer whether they consumed alcohol, tobacco/nicotine products and/or other drugs during pregnancy. The substances referred to in the questionnaire may have effects on brain and behavior development for a woman's offspring, this would be co-variable information. How much of a certain substance was used at the various phases of pregnancy can be calculated. This outcome is assessed at the post-class phase.
Change in Relationship Strength Levels as Measured by the Perceived Relationship Quality Components Inventory (PRQC) | Up to 12 months post birth
  Change in relationship strength level will be explored using the PRQC which will also be used to compare the MBCP group to the TAU group.
  The PRQC is an 18-item self-report questionnaire with three questions in each of the six constructs: satisfaction, commitment, intimacy, trust, passion, and love. Ratings are on a 7-point scale: 1-Not at all to 7-Extremely. Total possible range of scores is 18-126. Higher scores indicate higher level of relationship strength. This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).
Change in Quality of Life as Measured by the EQ-5D5L Questionnaire | Up to 12 months post birth
  Change in quality of life will be explored using the EQ-5D5L which will also be used to compare the MBCP group to the TAU group.
  The EQ-5D5L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. Participants select which statement best fits them on five dimensions in the descriptive module: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants then rate how good or bad their health is that day on a scale of 0 (worst health you can feel) through 100 (best health you could feel). This outcome is assessed at all phases except screening (pre-class, post-class, 1 month follow-up, 3 month follow-up, and 12 month follow-up).

SECONDARY OUTCOMES:
Infant Enjoyment and Mother-Infant Attachment Differences as Measured by the Puppet Task (Lab-TAB Task) | At 12 months post birth
  Infant enjoyment in response to social stimulation as well as mother-infant interaction will be explored using the puppet task from the Lab-TAB battery. The MBCP group will be compared to the TAU group.
  The episode begins with the appearance of the puppets from under the table and is divided into 5 trials for scoring. Variables to be coded: a) latency to joy, b) intensity of smiling, c) laughter, d) positive vocalizations, e) positive motor acts, f) latency to approach, g) engagement with toy, h) parent behavior, and i) baseline state. This outcome is assessed at the 12 month follow-up.
Infant Anger and Mother-Infant Attachment Differences as Measured by the Arm Restraint Task (Lab-TAB Task) | At 12 months post birth
  Infant anger in response to physical restraint as well as mother-infant interaction will be explored using the arm restraint task from the Lab-TAB battery. The MBCP group will be compared to the TAU group.
  The restraint episode begins, for scoring purposes, when child is no longer able to reach the toy. There are two 30-second trials, each of which is divided into six 5-second epochs. For each of the 12 epochs, a "1" mark on the coding sheet indicates that the specified behavior occurred, and "0" indicates that it did not. Variables to be coded: a) latency to anger response, b) latency to sadness response, c) intensity of struggle, d) intensity of facial anger, e) intensity of facial sadness, f) presence of bodily sadness, g) intensity of distress vocalizations, h) baseline state, i) effectiveness of parent, and j) engagement with toy. This outcome is assessed at the 12 month follow-up.
Infant Pleasure and Mother-Infant Attachment Differences as Measured by the Peek-A-Boo Task (Lab-TAB Task) | At 12 months post birth
  Infant pleasure in response to social stimulation as well as mother-infant interaction will be explored using the peek-a-boo task from the Lab-TAB battery. The MBCP group will be compared to the TAU group.
  The episode begins with the first "Where's Mommy?" and consists of 6 trials, each one beginning with "Where's Mommy?" and ending with the beginning of the next "Where's Mommy?," except for the last trial that ends 15 s after it begins. The trials are coded by indicating the occurrence of the specified behavior, or by rating the intensity of the behavior. When an intensity rating is requested, the highest intensity observed should be coded. Variables to be coded: a) latency to joy, b) intensity of smiling, c) laughter, d) positive vocalization, e) positive motor activity, f) effectiveness of parent, and g) baseline state. This outcome is assessed at the 12 month follow-up.
Emotion Regulation and Mother-Infant Attachment Differences as Measured by the Strange Situation | At 12 months post birth
  Infant social-emotional skills, such as emotion regulation, as well as mother-infant interaction will be explored using the Strange Situation. The MBCP group will be compared to the TAU group.
  In the Strange Situation, the observer notes down the behavior displayed during 15-second intervals and scores the behavior for intensity on a scale of 1 to 7. Attachment styles are based primarily on 4 interaction behaviors: proximity and contact seeking, contact maintaining, avoidance of proximity and contact, and resistance to contact and comforting. Other behaviors observed include exploratory behaviors, search behaviors and affect displays. This outcome is assessed at the 12 month follow-up.
Brain Structure and Functional Connectivity Differences as Measured by Magnetic Resonance Imaging (MRI) Scans | At 1 month post birth
  Brain structure and functional connectivity during resting state and task state will be explored using MRI techniques. The MBCP group will be compared to the TAU group.
  The brain areas of particular interest is the amygdala and relevant cortico-limbic areas. This outcome is assessed at the 1 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Duncan, PhD, Principal Investigator — Center for Healthy Minds; Sarah Short, PhD, Principal Investigator — Center for Healthy Minds
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected as part of the study may be shared with other researchers upon request or shared publicly in an open science format. Other researchers within and outside of UW-Madison may request to use data from this study. Data may be shared as Supplemental Information uploaded to a journal website and/or shared on a UW data sharing website.
Time Frame: Data will be available after data collection is complete. The time frame has not been set yet.
Access Criteria: Any future research utilizing these data will be submitted as a separate application to the Institutional Review Board prior to their use, if required by IRB policies and/or guidance. Researchers within and outside UW-Madison may request access to data.